CLINICAL TRIAL: NCT03088566
Title: Implementation of the D-Foot at the Department of Prosthetics and Orthotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Hellstrand Tang, Certified prosthetist and orthotist, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 224651
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Randomised controlled study. One group will be foot screened following the routine described in the web program, the D-Foot. The other group will be foot screened by the use of conventional methods.
Who Masked: Participant
Masking Description: The randomisation will be determined by sequencing patients into on of the two groups following the grouping found in closed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The D-Foot method (Experimental): The patients are being foot screened following the routine that is programmed in the D-Foot.
  Interventions: Procedure: The D-Foot method
- Conventional foot screening (Active Comparator): The patients are being foot screened according to conventional methods.
  Interventions: Procedure: Conventional foot screening

INTERVENTIONS:
Procedure: The D-Foot method — The D-Foot method is a standardised routine of foot screening. The D-Foot i web program aimed to be used on a surf plate.
  Arms: The D-Foot method
Procedure: Conventional foot screening — The foot screening is performed with clinical conventional methods.
  Arms: Conventional foot screening

SUMMARY:
Early identification of potential risk factors for the onset of diabetic foot ulcers are recommended. However, in a Swedish context, there has been no standardised routines to be used in the foot screening procedure. In this study a new standardised routine, the D-Foot, will be tested at the Department of Prosthetics and Orthotics. The usability of the web program will be tested.

DETAILED DESCRIPTION:
The primary research questions are"how do patients with diabetes perceive the foot screening?" and "do the perception differ in the group that was foot screened by the use of the D-Foot compared to the group that was foot screened with conventional methods?"

ELIGIBILITY:
Inclusion Criteria:

* diabetes
* patients referred to the Department of Prosthetics and Orthotics at Sahlgrenska University Hospital with the aim to be provided with assistive devices with the purpose to protect the feet from foot ulcers
* be able to read and understand the Swedish language

Exclusion Criteria:

*being unable to read and understand the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 111 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patients reported experience measure (PREM) | one month
  Orthotic and Prosthetic Users survey will be used to evaluate if the PREM scores are higher in the group that was foot screened following the D-Foot method. MEASURE is scored to range from 0 (the lowest possible score) to 100 (the highest possible score).
Patients reported experience measure (PREM) | one month
  A selection of questions from the Swedish national patient survey will be used to evaluate if the PREM scores are higher in the group that was foot screened following the D-Foot method

SECONDARY OUTCOMES:
PREM | one month
  The system usability scale will be used to calculate the level of usability among the patients that were randomized to the D-Foot group
Patients reported outcome measure (PROM) | one month
  The answers from the EQ-5D will be used to describe the health related quality of life of the study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prostetics & Orthotics, Gothenburg, Region Västragötaland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hellstrand Tang U, Tranberg R, Sundberg L, Scandurra I. How do patients and healthcare professionals experience foot examinations in diabetes care? - A randomised controlled study of digital foot examinations versus traditional foot examinations. BMC Health Serv Res. 2024 Nov 12;24(1):1387. doi: 10.1186/s12913-024-11674-w. PMID 39533310